CLINICAL TRIAL: NCT05082545
Title: A Phase I Clinical Study on the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of SHR-2002 Injection in Combination With SHR-1316 in Patients With Advanced Malignant Tumors
Brief Title: Phase I Study of SHR-2002 + SHR-1316 in Patients With Advanced Malignant Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-2002-102; SHR-2002-I-102 (Other: Jiangsu Hengrui Pharmaceuticals Ltd.)
Record Dates: First submitted 2021-09-15; First posted 2021-10-19 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2023-12

CONDITIONS: Advanced Malignant Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose escalation:SHR-2002+SHR-1316 (Experimental): SHR-2002 +SHR-1316 C1D1 SHR-2002,C1D22 SHR-2002+SHR-1316, C2 SHR-2002+SHR-1316
  Interventions: Drug: SHR-2002 and SHR-1316
- Dose expansion stage: SHR-2002+SHR-1316 (Experimental): Dose expansion of SHR-2002 will be decided after finishing few cohorts in Dose escalation part.
  Interventions: Drug: SHR-2002 and SHR-1316
- Indication expansion stage：SHR-2002+SHR-1316 (Experimental): Indication expansion of SHR-2002 will be decided after finishing few cohorts in Dose expansion part.
  Interventions: Drug: SHR-2002 and SHR-1316

INTERVENTIONS:
Drug: SHR-2002 and SHR-1316 — Cohort study

SUMMARY:
This is Phase 1 study FIH to check "Dose Escalation, Dose expansion and Indication expansion". This study is AUSTRALIA only study.

ELIGIBILITY:
Subjects must meet all the following criteria to be eligible for enrollment into the study:

1. Ability to understand and voluntarily agrees to participate by giving written informed consent for the study;
2. Male or female aged ≥18 years at the time of signing the ICF;
3. Histopathologically or cytologically documented advanced or metastatic malignancies and failed or intolerable to previous standard therapy, has no available standard of care therapy or refused standard therapy;
4. An Eastern Cooperative Oncology Group (ECOG) performance status (PS) score of 0 or 1 (Appendix 2);
5. Female and male patients of reproductive potential must agree to use highly effective contraception during the study treatment period and within 6 months after the last investigational drug administration.

Subjects who meet any of the following criteria will be excluded from the study:

1. Patients with known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
2. Patients with tumor-related pain that cannot be controlled as determined by the investigator.
3. Systemic anti-tumor therapy within 28 days prior to the first dose of the study treatment
4. History of autoimmune diseases, except for Type 1 diabetes (blood glucose can be controlled by insulin therapy)
5. History of clinically significant cardiovascular or cerebrovascular diseases within 6 months prior to the first dose of study treatment.
6. Known history of serious allergic reactions to the investigational product or its main ingredients;
7. History of immunodeficiency, including positive HIV serum test result and other acquired or congenital immunodeficiency diseases, or history of organ transplantation;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2023-07-17 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
Adverse events | Screening up to study completion, an average of 2 years
  Number of subjects with adverse events (AEs)
Number of participants experiencing Dose-Limiting Toxicities (DLTs) | Up to 42 days
  According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE v.5.0)

SECONDARY OUTCOMES:
PK of SHR-2002 + SHR-1316 | Before and after SHR-2002 and SHR-1316 infusion throughout the study, an average of 2 years
  To check Maximum concentration (Cmax)
PK of SHR-2002 + SHR-1316 | Before and after SHR-2002 and SHR-1316 infusion throughout the study, an average of 2 years
  To check AUC last
Immunogenicity of SHR-2002 + SHR-1316 | Before and after SHR-2002 and SHR-1316 infusion throughout the study, an average of 2 years
  ADA of SHR-2002 + SHR-1316

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (4):
  - Icon Cancer Centre, Brisbane, Queensland
  - Linear clinical research, Perth, Western Australia
  - Scientia Clinical research, Sydney
  - Liverpool Hospital, Sydney